CLINICAL TRIAL: NCT06071871
Title: A Phase II Trial of Polatuzumab Vedotin, Obinutuzumab and Glofitamab As a Peri-CAR-T Cell Treatment Strategy in Large B-cell Lymphoma
Brief Title: A Trial of Polatuzumab Vedotin, Obinutuzumab and Glofitamab As a Peri-CAR-T Cell Treatment Strategy in Large B-cell Lymphoma
Acronym: PORTAL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/150862; 2022-003727-17 (EudraCT Number)
Record Dates: First submitted 2023-08-23; First posted 2023-10-10 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Large B-cell Lymphoma
Keywords: Glofitamab; Polatuzumab vedotin; Obinutuzumab; Bridging therapy; Large B-cell Lymphoma
MeSH Terms: interventions — glofitamab; polatuzumab vedotin; obinutuzumab

STUDY DESIGN:
Intervention Model Description: Part 1: 42 patients, Part 2: 42-57 patients (some Part 1 patients may also participate in Part 2)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part 1 (Experimental): Patients whose large B-cell lymphoma has progressed/not responded to previous treatment and are due to start standard CAR-T therapy.
  All patients receive 2 cycles of glofitamab and polatuzumab vedotin (Glofit-Pola). Obinutuzumab pre-treatment is given on cycle 1 day 1.
  Patients have a PET-CT scan to check the response after cycle 2. If the scan shows a response and patients are still suitable for CAR-T cell therapy, patients will proceed to receive planned CAR-T therapy and will not receive further Glofit-Pola in Part 1. If not, patients can receive 4 more cycles of glofitamab and polatuzumab vedotin, and then 6 cycles of glofitamab.
  Interventions: Drug: Glofitamab; Drug: Polatuzumab vedotin; Drug: Obinutuzumab
- Part 2 (Experimental): Patients whose large B-cell lymphoma has progressed/not responded after standard CAR-T cell therapy.
  All patients receive 6 cycles of glofitamab and polatuzumab vedotin (Glofit-Pola), and then 6 cycles of glofitamab alone. Obinutuzumab pre-treatment is given on cycle 1 day 1.
  Interventions: Drug: Glofitamab; Drug: Polatuzumab vedotin; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Glofitamab — Glofitamab is given intravenously at a dose of 2.5mg over 4 hours on Cycle 1 Day 8. Patients need to stay in hospital for 24 hours.
  Glofitamab is given intravenously at a dose of 10mg over 2 hours on Cycle 1 Day 15. (Patients may need to stay in hospital for 24 hours.) Glofitamab is given intravenously at a dose of 30mg over 2 hours on Day 1 of Cycles 2-12 (as relevant).
  Other Names: Columvi
Drug: Polatuzumab vedotin — Polatuzumab is given intravenously at a dose of 1.8mg/kg on Cycle 1 Day 2, and then Day 1 of Cycle 2-Cycle 6.
  Other Names: Polivy
Drug: Obinutuzumab — Obinutuzumab pre-treatment is given intravenously at a dose of 1g on Cycle 1 Day 1.
  Other Names: Gazyvaro

SUMMARY:
The PORTAL study will test a new combination of drugs (glofitamab, polatuzumab vedotin and obinutuzumab) in patients with large B-cell lymphoma (LBCL) that has come back (relapsed) or not responded to previous treatment. It will determine how safe and effective the combination of these cancer drugs is in treating LBCL before and after CAR-T cell therapy.

DETAILED DESCRIPTION:
This is a phase 2, open label trial conducted in 2 parts.

The overall aim is:

Part 1: To determine the efficacy of Pola-Glofit as bridging treatment to CAR-T cell therapy in patients with relapsed or refractory large B cell lymphomas.

Part 2: To determine the efficacy of Pola-Glofit in patients with relapsed or refractory large B cell lymphomas who have failed to achieve CMR, or progressed after CAR-T cell therapy.

Treatment consists of:

Part 1: Patients will receive 2 cycles of Pola-Glofit. Obinutuzumab is given 7 days before the first dose of Glofit. After 2 cycles, patients have a PET-CT scan to check the response. If the scan shows a response and the patient is still suitable for CAR-T, patients will receive planned CAR-T therapy. If the patient is not suitable to continue with CAR-T, patients can receive up to 4 more cycles of Pola-Glofit, and then 6 cycles of Glofit.

Part 2: Patients will receive 6 cycles of Pola-Glofit, and then 6 cycles of Glofit. Obinutuzumab is given 7 days before the first dose of Glofit.

For both Part 1 and Part 2, all cycles are 21 days. A step-up dosing regimen will be followed:

* Cycle 1 Day 1: Obinutuzumab is given intravenously at a dose of 1g over 4-5 hours.
* Cycle 1 Day 2: Polatuzumab is given intravenously at a dose of 1.8mg/kg over 90 minutes.
* Cycle 1 Day 8: Glofitamab is given intravenously at a dose of 2.5mg over 4 hours. Patients need to stay in hospital for 24 hours.
* Cycle 1 Day 15: Glofitamab is given intravenously at a dose of 10mg over 2 hours. (Patients may need to stay in hospital for 24 hours.)
* From Cycle 2-6, Polatuzumab is given intravenously at a dose of 1.8mg/kg over 30 minutes on Day 1, and Glofitamab is given intravenously at a dose of 30mg over 2 hours on Day 1.
* From Cycle 7-12, Glofitamab is given intravenously at a dose of 30mg over 2 hours on Day 1.

Patients will be followed up until the last patient completes their 1 year post-treatment follow up visit.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven CD20+ LBCL (with CD20 positivity at any timepoint) including diffuse large B cell lymphoma, high grade B cell lymphoma with MYC, BCL2 and/or BCL6 (double/triple hit lymphoma), high grade B cell lymphoma not otherwise specified (NOS), primary mediastinal B-cell lymphoma or transformed follicular lymphoma.

  * Part 1: Relapsed or refractory disease and eligible for CAR T-cell therapy in the UK and in need of systemic bridging in the opinion of the local investigator.
  * Part 2: Failed to achieve CMR (Deauville score 1-3) on PET scan 1-month post CAR-T or progressed at any point post CAR-T (patients in part 2 may have been previously enrolled in Part 1 and responded to Pola-Glofit bridging or be de novo patients who are naïve to this combination)
* At least one measurable target lesion
* Patient has recent archival biopsy tissue available or is willing to undergo a new biopsy.
* ECOG performance status:

  * Part 1: ECOG PS 0/1
  * Part 2: ECOG PS 0-2
* Life expectancy of ≥ 12 weeks
* Adequate haematological status.
* Adequate liver and renal function
* Negative test for hepatitis B, hepatitis C, HIV and SARS-CoV-2

Exclusion Criteria:

* Patients with known active infection
* Current ≥ Grade 2 peripheral neuropathy
* History of confirmed progressive multifocal leukoencephalopathy
* Current evidence of CNS lymphoma
* Patients with another invasive malignancy in the last 2 years
* Significant history of cardiovascular disease
* Active autoimmune disease or immune deficiency
* Severe neurological disorder
* Uncontrolled tumour-related pain
* Uncontrolled pleural effusion, pericardial effusion, or ascites
* Treatment with other standard anti-cancer radiotherapy/chemotherapy including investigational therapy and targeted therapy within 4 weeks prior to cycle 1 day 1
* Prior solid organ transplantation
* Prior allogeneic stem cell transplant
* Autologous SCT within 100 days prior to cycle 1 day 1
* Any history of immune related ≥ Grade 3 adverse events
* Ongoing corticosteroid use > 25 mg/day of prednisone or equivalent within 4 weeks prior to study treatment
* Treatment with systemic immunosuppressive medication within 2 weeks prior to initiation of study treatment
* Administration of a live, attenuated vaccine within 4 weeks prior to cycle 1 day 1
* History of severe allergic anaphylactic reactions to chimeric or humanised monoclonal antibodies or recombinant antibody-related fusion proteins.
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the obinutuzumab, polatuzumab vedotin and/or glofitamab formulation.
* Known or suspected history of HLH

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Part 1: Overall Response Rate (ORR) to Pola-Glofit as bridging prior to CAR-T cell infusion | At Cycle 2 Day 14-19 (or earlier) (each cycle is 21 days)
  To determine the efficacy of Pola-Glofit as bridging treatment to CAR-T cell therapy in patients with r/r LBCL.
  ORR i.e. the proportion of patients achieving response (Complete Metabolic Response or Partial Metabolic Response) after Pola-Glofit bridging but prior to CAR-T cell infusion, assessed by central review as per 2014 Lugano Classification. This will be presented as a rate with a 70% confidence interval.
Part 2: Progression Free Survival (PFS) at 6 months | From the date of registration at Part 2 until the date of first disease progression or death, whichever comes first, assessed up to 4 years
  To determine the efficacy of Pola-Glofit in patients with LBCL who have failed to achieve CMR, or progressed after CAR-T cell therapy.
  PFS at 6 months will be analysed using Kaplan-Meier survival analysis, with the rate at 6 months (with 70% CI) presented. The median (if reached) and plot will also be given.

SECONDARY OUTCOMES:
Part 1: Complete Metabolic Response (CMR) rate to Pola-Glofit as bridging prior to CAR-T cell infusion | At Cycle 2 Day 14-19 of bridging treatment (each cycle is 21 days)
  Per Lugano 2014 criteria
Part 1: Overall Survival (OS) and Progression Free Survival (PFS) | From the date of registration at Part 1 until the date of disease progression or death (PFS), or death (OS). This will be assessed from the date of registration until up to 4 years.
  Medians (if reached), rates at 6 months and 1 year and plots will be presented
Part 1: Safety and toxicity of Pola-Glofit as bridging therapy | From registration and during Part 1 bridging treatment, until end of post-treatment safety reporting window (up to six months after last dose of obinutuzumab, plus a further 35 days after last dose of polatuzumab vedotin or last dose of glofitamab)
  Assessed by CTCAE criteria v5 and ASTCT 2019 criteria for CRS/ICANS adverse events. Assessed in all patients given at least one dose of study treatment in part 1.
Part 1: CAR-T associated toxicity post Pola-Glofit bridging following CAR-T therapy | Between Day 0 and Day 28 following CAR-T therapy
  Assessed in all patients given at least one dose of study treatment in part 1 and infused. Assessed by CTCAE criteria v5 and ASTCT 2019 criteria for CRS/ICANS adverse events.
Part 1: Response rate post CAR-T for all infused patients | From CAR-T infusion until 6 months post CAR-T therapy
  Per Lugano 2014 criteria. Response rates at 1, 3 and 6 months post CAR-T therapy.
Part 1: Duration of Response (DoR) and Duration of Complete Response (DoCR) for Pola-Glofit and CAR-T | From the date of first response until disease progression. This will be assessed from the date of registration until up to 4 years.
  Response defined as PR (partial response) or better.
Part 1: Non-Relapse Mortality (NRM) | From the date of registration until the date of NRM. This will be assessed from the date of registration until up to 4 years.
  NRM rates at 6 months and 1 year
Part 2: Complete Metabolic Response (CMR) rate to Pola-Glofit/Glofitamab at any point | From the date of registration until up to 4 years
  Per Lugano 2014 criteria
Part 2: Response rate for patients who received Pola-Glofit bridging versus those who have not | From the date of registration until Cycle 5 (approximately 12 weeks. Each cycle is 21 days).
  Per Lugano 2014 criteria. Response rates following 2 and 5 cycles of Part 2 treatment.
Part 2: Safety and toxicity of Pola-Glofit post CAR-T therapy | Throughout Part 2 treatment until end of post-treatment safety reporting window (up to six months after last dose of obinutuzumab, plus a further 35 days after last dose of polatuzumab vedotin or last dose of glofitamab)
  Assessed by CTCAE criteria v5 and ASTCT 2019 criteria for CRS/ICANS adverse events. Assessed in all patients given at least one dose of study treatment in part 2.
Part 2: Overall Survival (OS) | From the date of registration for Part 2 until the date of death, assessed up to 4 years.
  Median (if reached), rates at 6 months and 1 year (with 95% CIs) and plots will be presented.
Part 2: Duration of Response (DoR) | From the date of first response until disease progression, assessed up to 4 years.
  Response defined as PMR (partial metabolic response) or better.
Part 2: Duration of Complete Response (DoCR) | From the date of first complete metabolic response (CMR) until disease progression, assessed up to 4 years.
Part 2: Non-Relapse Mortality (NRM) | NRM will be measured from the date of registration until the date of NRM. This will be assessed from the date of registration until up to 4 years. NRM rates will be presented at 6 months and 1 year.
  NRM rates will be presented at 6 months and 1 year.
Part 2: Progression Free Survival (PFS) (at 12 months) | PSF will be measured from the date of registration at Part 2 until the date of disease progression. This will be assessed from the date of registration until up to 4 years. The median rate at 12 months will be presented.
  Median (if reached), rate at 12 months (with 95% CI) and plot will be presented

CONTACTS AND LOCATIONS:
Overall Officials: William Townsend, Principal Investigator — University College London Hospitals
Locations (5):
- United Kingdom (5):
  - Kings College Hospital NHS Foundation Trust, London
  - University College London Hospitals NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No